CLINICAL TRIAL: NCT05660785
Title: The Efficacy and Safety of Herombopag Combined With Cyclosporine for Patients With Non Severe Aplastic Anemia
Brief Title: Herombopag Added to Cyclosporine in Non Severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022049
Record Dates: First submitted 2022-11-23; First posted 2022-12-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-01

CONDITIONS: Non Severe Aplastic Anemia; Untreated
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CsA + Herombopag (Experimental): Herombopag combined with cyclosporine
  Interventions: Drug: Herombopag

INTERVENTIONS:
Drug: Herombopag — Hetrombopag is a TPO receptor agonist approved in China in 2021 for idiopathic thrombocytopenic purpura (ITP) and second-line severe aplastic anemia (SAA). Indications of chemotherapy-induced thrombocytopenia (CIT), pediatric/juvenile ITP and naive severe aplastic anemia are under development. Hetrombopag was granted Orphan Drug Designation by FDA for the treatment of CIT.
  Cyclosporine A is a calcineurin inhibitor, which has an effect on reducing T-cell proliferation and activation, can reverse pancytopenia and alleviate transfusion requirements in NSAA.
  Other Names: Cyclosporine A

SUMMARY:
This is a prospective, multicenter, single-arm, phase 2 trial. The aim of this study is to evaluate the efficacy and safety of herombopag combined with cyclosporine for patients with non severe aplastic anemia (NSAA).

DETAILED DESCRIPTION:
This study aims to improve the 24 weeks response rate. The sample size is calculated based on Simon's two-stage design. The first stage of the study enrolled a cohort of 15 patients. If after 24 weeks at least 9 patients achieved a response, then enrollment was expanded to a total of 43 patients. The null hypothesis was unaccepted if more than 26 of 43 patients achieved the response. Accounting for a 20% dropout rate, the estimated final sample size was 54 patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with the requirements for this study and written informed consent.
* Male or female age ≥ 18 years
* Diagnosis of untreated non severe aplastic anemia.
* Platelet counts < 50 x 10^9/L at least 2 times consecutively (time interval ≥ 1 week)

Exclusion Criteria:

* Receive immunosuppressive therapy more than 4 weeks before enrollment
* Treatment with TPO-RA within 1 week before enrollment
* Inherited bone marrow failure syndromes
* Bone marrow fibrosis grade ≥ 2
* The presence of hemolytic PNH clone
* The presence of clonal karyotypic abnormalities (del(20q), +8 and -Y are not included in this category)
* Previously treated with TPO-RA ≥ 4 weeks
* Previously received immunosuppressive therapy ≥ 12 weeks
* Ferritin > 1000 ng/ml (The increased level of Ferritin led by infection is not included in this category)
* Have an allergy to eltrombopag or any other part of this medicine.
* History of radiotherapy and chemotherapy for malignant solid tumors
* Cytopenia caused by other non-hematologic diseases, including liver cirrhosis, active rheumatic connective tissue disease, and persistence of infectious diseases, etc
* Abnormal liver function: ALT or AST > 3 ULN, or TBil > 1.5 ULN after treatment.
* Abnormal kidney function: Creatinine clearance < 30 ml/min, or serum creatinine (sCr) >1.5 ULN
* Patients with diabetic nephropathy, neuropathy, or eye disease
* Patients with poorly controlled hypertension or cardiac arrhythmia
* Patients with congestive heart failure and the NYHA grade ≥ 3 historically or currently, and LVEF < 45% within 4 weeks before enrollment
* History of arteriovenous thrombosis within 1 year before enrollment
* Participation in another clinical trial within 4 months before the start of this trial
* Pregnant or breast-feeding patients
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 24 weeks
  Percentage of patients with hematological response. Hematological response is evaluated by hemoglobin, platelet and neutrophil count in the routine blood test.

SECONDARY OUTCOMES:
Robust response rate | 24 weeks
  Percentage of patients with robust response, including complete response, near complete response, very good partial response(VGPR) and Meaningful partial response(mPR). These are evaluated by hemoglobin, platelet and neutrophil count in the routine blood test.
Proportion of patients with abnormal karyotype changes | Baseline and 24 weeks
  The abnormal karyotype was examined by karyotype test
Time duration for patients achieving hematological response | A minimum of 2 years of planned follow-up
  Duration time was calculated from response to relapse.
Change of the health-related quality of life | Baseline and 24 weeks
  Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) is used to assess the health-related quality of life of patients. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
Incidence of the adverse event | 24 weeks
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event.
Severity of the adverse event | 24 weeks
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the severity.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Tangshan Central Hospital, Tangshan, Hebei
  - Zhoukou Central Hospital, Zhoukou, Henan
  - The Second Affilated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Regenerative Medicine Center, Tianjin, Tianjin Municipality